CLINICAL TRIAL: NCT04034849
Title: Effects of Photobiomodulation With Low-Level Laser Therapy in Burning Mouth Syndrome: A Randomized Clinical Trial
Brief Title: Effects of Photobiomodulation in Burning Mouth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosa María López-Pintor Muñoz (Other)
Responsible Party: Sponsor-Investigator, Rosa María López-Pintor Muñoz, Associate Professor; Co-director Speciality in Oral Medicine, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0003
Record Dates: First submitted 2019-07-19; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Burning Mouth Syndrome
Keywords: Low-level Laser Therapy; Burning Mouth Syndrome; Photobiomodulation; Visual Analogue Scale; Oral Health Impact Profile; Clinical Trial
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized single blind placebo controlled study
Who Masked: Participant
Masking Description: All patients were masked during all the trial. They wore protective glasses and were also advised to close their eyes during treatment. In addition, the laser was programmed not to emit any type of sound alarm. One clinician collected the Visual Analogue Scale and the questionnaires fulfilled by the patients and another clinician applied the laser treatment. All patients were warned of not speaking with the laser clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Low-Level Laser Therapy was applied in the test group with a Diode Laser Fox (A.R.C. Laser, Italy) using these parameters: a wavelength of 810 nm, a power of 0.6 W, a power density of 1.2 W/cm2, a beam area of 0.08 cm2 and an energy of 6 J with an application time per point of 10 seconds in 56 points (3 in the vestibular mucosa of the 4 quadrants, 6 in each of the two buccal mucosa, 6 in the hard palate, 4 in each lateral of the tongue, 6 in the dorsum of the tongue and 4 sublingual points) with a distance between points of 2mm. It was applied, therefore, a dose of 12 J/cm2 in a continuous mode in a total of 10 sessions, 2 sessions per week for 5 weeks.
  Interventions: Radiation: Photobiomodulation
- Placebo group (Placebo Comparator): Low-Level Laser Therapy was applied in the placebo group with a Diode Laser Fox (A.R.C. Laser, Italy) turned off with an application time per point of 10 seconds in 56 points (3 in the vestibular mucosa of the 4 quadrants, 6 in each of the two buccal mucosa, 6 in the hard palate, 4 in each lateral of the tongue, 6 in the dorsum of the tongue and 4 sublingual points) with a distance between points of 2mm. It was applied, therefore, a dose of 12 J/cm2 in a continuous mode in a total of 10 sessions, 2 sessions per week for 5 weeks.
  Interventions: Radiation: Placebo

INTERVENTIONS:
Radiation: Photobiomodulation — Photobiomodulation whit Low-Level Laser Therapy
  Arms: Test group
Radiation: Placebo — Device turned off
  Arms: Placebo group

SUMMARY:
The main objective of this study is to assess the effects of Photobiomodulation with Low-level Laser Therapy to the pain management in Burning Mouth Syndrome patients, besides assessing their impact on the different aspects of their quality of life, using the necessary questionnaires to evaluate all the outcomes of chronic pain.

DETAILED DESCRIPTION:
Study design A randomized, single blind, clinical trial was performed among patients with Burning Mouth Syndrome who attended the Oral Medicine Specialist Degree Program at the School of Dentistry at Complutense University in Madrid. This study was approved by the Hospital San Carlos Ethics Committee in Madrid (IEC no. 17/311-R_P) according with the principles of the Helsinki Declaration. This clinical study followed the guidelines established by the Consort Statement (http://www.consort-statement.org/).

Participants Adult patients older than 18 years of age who fulfilled the International Classification of Headache Disorders (ICHD-3) diagnostic criteria for BMS were consecutively included in this study. Patients not interested in participate in the study, unable to understand or answer the questionnaires and follow the appointments, patients suffering hiposialia or Sjögren's syndrome, patients who had received head and neck radiotherapy, pregnant women, patients with uncontrolled systemic diseases (diabetes, thyroid diseases, fibromyalgia or anemia) and patients suffering burning mouth symptoms secondary to local factors were excluded. Patients also had to read and sign and informed consent prior to inclusion in the study.

Before beginning the treatment, all patients provided a full medical history and a complete blood test including blood levels of iron, vitamin B12, folic acid, TSH and basal glucose levels. Patients who did not provide the blood tests, did not attend any of the appointments or follow-ups or did not fulfill correctly the questionnaires were removed from the study.

Interventions LLLT was applied in the study group with a Diode Laser Fox (A.R.C. Laser, Italy) using these parameters: a wavelength of 810 nm, a power of 0.6 W, a power density of 1.2 W/cm2, a beam area of 0.08 cm2 and an energy of 6 J with an application time per point of 10 seconds in 56 points (3 in the vestibular mucosa of the 4 quadrants, 6 in each of the two buccal mucosa, 6 in the hard palate, 4 in each lateral of the tongue, 6 in the dorse of the tongue and 4 sublingual points) with a distance between points of 2mm. It was applied, therefore, a dose of 12 J/cm2 in a continuous mode in a total of 10 sessions, 2 sessions per week for 5 weeks. The laser was applied perpendicularly in contact with the mucosa. All patients and the clinician wore the protective eyeglasses provided with the laser device.

For the placebo group the Low-Level Laser Therapy was applied in the same 56 points, 10 seconds per point and the same number of sessions but with the device turned off.

Outcomes Medical reports, medical questionnaires and blood tests (iron, vit B12, folic acid, TSH and basal glucose) were collected before starting the laser application. Pain was assessed using a Visual Analogue Scale (0-10 cm) by the patients before starting each session and at two follow-up sessions, 1 and 4 months after finishing the treatment.

Different questionnaires validated to Spanish were also fulfilled by patients. The questionnaires were the Short Form 36 Health Survey (SF-36) for the general health status, the Oral Health Impact Profile (OHIP-14) for the oral patient's quality of life, the Epworth sleepiness scale, the psychometric test Symptom Check List 90 (SCL 90), the Beck's depression inventory and the McGill Pain Questionnaire. These questionnaires were fulfilled baseline and at the end of the 10 laser sessions and in the 1st and 4th-months follow-ups.

Sample size The sample size was calculated considering the previous study performed by Sikora et al, 2018 applying Low-Level Laser Therapy in similar parameters with a placebo group. We considered that the acceptable improvement in Laser group would be 4 points in VAS for pain. With a p = 0.05, a statistical power of 90% to detect this difference would require 10 subjects in each study group.

Randomization Burning Mouth Syndrome patients were randomly assigned to one of the treatments (Low-Level Laser Therapy or placebo) in a 1:1 ratio using a computer-generated algorithm stratified by using a block sized of 4. The patient's arrival number was his assigned number for the study following a correlative sequence. Group assignation for each number was kept in a sealed envelope that was no opened until the moment of treatment. An investigator not involved in the Low-Level Laser Therapy performed the randomization. The clinician who applied the Low-Level Laser Therapy was not involved in this process.

Blinding All patients were blinded during all the trial. They wore protective glasses and were also advised to close their eyes during treatment. In addition, the laser was programmed not to emit any type of sound alarm. One clinician collected the VAS and the questionnaires fulfilled by the patients and another clinician applied the laser treatment. All patients were warned of not speaking with the laser clinician. Blinding was revealed after all participants finished the trial, and all the data were analyzed

Statistical methods All the analysis was done using SPSS version 25.0 (SPSS Inc. New York, NY, USA). Statistical analysis included basic descriptive statistics. Comparison of categorical variables was done using chi-square or Fisher's exact test and comparison of continuous variables between test and placebo groups was done using Mann-Whitney U test. Wilcoxon signed-rank test was used to determine whether the intragroup decreases in the different questionnaires were statistically significant. Differences were considered significant if p was less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who fulfilled the International Classification of Headache Disorders (ICHD-3) diagnostic criteria for Burning Mouth Syndrome Exclusion Criteria
* Patients not interested in participate in the study, unable to understand or answer the questionnaires and follow the appointments, patients suffering hiposialia or Sjögren's syndrome, patients who had received head and neck radiotherapy, pregnant women, patients with uncontrolled systemic diseases (diabetes, thyroid diseases, fibromyalgia or anemia) and patients suffering burning mouth symptoms secondary to local factors

Ages: 31 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analogue Scale for Pain | Baseline (day 1), Session2 (day 4), Session 3 (day 8), Session 4 (day 11), Session 5 (day 15), Session 6 (day 18), Session 7 (day 22), Session 8 (day 25), Session 9 (day 29), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up(day 150)
  Pain was assessed using a Visual Analogue Scale (0-10 cm) by the patients before starting each session and at two follow-up sessions, 1 and 4 months after finishing the treatment.

SECONDARY OUTCOMES:
Description of Pain: Mc Gill Pain Questionnaire validated to Spanish | Baseline (day 1), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up (day 150)
  The patient is provided with a form comprising instructions and 20 word groups. The patient is instructed to read each word group and decide whether there is a work in the group which describes the pain he/she is experiencing there and then. The patient should circle one word in the group, which describes their pain. If there is no word in the group, which describes their pain, they are to move on to the next group until they have completed each of the 20 groups.
  Groups 1 to 10 are words used to describe sensory experience, groups 11 to 15 are affective words, 16 is evaluative and 17 to 20 are miscellaneous groups.
General Health Short Form with the 36 Health Survery validated to Spanish | Baseline (day 1), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up (day 150)
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health
Oral patient's quality of life with the Oral Health Impact Profile 14 validated to Spanish | Baseline (day 1), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up (day 150)
  This questionnaire includes 14 questions about oral pain, physical, psychological, and social limitations and disabilities whose score range from 0 to 4. The total score varies from 0 to 56. Poorer scores correspond to low quality of life.
Epworth sleepiness scale validated to Spanish | Baseline (day 1), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up (day 150)
  The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates that expert medical advice should be sought. For instance, scores of 11-15 are shown to indicate the possibility of mild to moderate sleep apnea, where a score of 16 and above indicates the possibility of severe sleep apnea or narcolepsy.
Psychometris test Symptom Check List 90 validated to Spanish | Baseline (day 1), Session 10 (day 32), 1st month follow-up (day 60), 4th month follow-up (day 150)
  According to the overview given by the publisher, the SCL-90-R is normed on individuals 13 years and older. It consists of 90 items with options from 0 to 4 and takes 12-15 minutes to administer, yielding nine scores along primary symptom dimensions and three scores among global distress indices. The primary symptom dimensions that are assessed are somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, and a category of "additional items" which helps clinicians assess other aspect of the clients symptoms (e.g. item 19, "poor appetite"). The three indices are global wellness index, hardiness, and symptom free. The higher scores, the poorer psychological status.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa María López-Pintor, PhD, Study Director — Universidad Complutense Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Montero-Martin J, Bravo-Perez M, Albaladejo-Martinez A, Hernandez-Martin LA, Rosel-Gallardo EM. Validation the Oral Health Impact Profile (OHIP-14sp) for adults in Spain. Med Oral Patol Oral Cir Bucal. 2009 Jan 1;14(1):E44-50. PMID 19114956